CLINICAL TRIAL: NCT05631379
Title: Influence of Body Composition, Nutritional Status and Inflammatory Markers on Survival and Postoperative Outcome in Patients Operated on for Primary Retroperitoneal Sarcoma: Report From Institute of Oncology Ljubljana
Brief Title: Influence of Nutritional Status on Oncologic and Operative Outcome in Patients Operated for Retroperitoneal Sarcoma
Status: Completed | Type: Observational
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: ERID-KSOPKR-0081/2020
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Retroperitoneal Sarcoma; Body Composition; Malnutrition; Sarcopenia; Sarcopenic Obesity; Myosteatosis
MeSH Terms: conditions — Malnutrition; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- All patients meeting inclusion criteria: All patients meeting inclusion criteria
  Interventions: Diagnostic Test: GLIM malnutrition criteria; Diagnostic Test: Prognostic Nutritional Index (PNI); Diagnostic Test: The high-sensitivity modified Glasgow prognostic score
- Subgroup of patients with available preoperative CT/MRI scans: Subgroup of patients with available preoperative CT/MRI scans will be detected and body composition measurements will be assessed min order to detect nutrition-related syndromes
  Interventions: Other: Measurement of body composition with computed tomography (CT); Diagnostic Test: GLIM malnutrition criteria; Diagnostic Test: EWGSOP2 sarcopenia criteria; Diagnostic Test: ESPEN-EASO criteria for sarcopenic obesity; Diagnostic Test: Prognostic Nutritional Index (PNI); Diagnostic Test: The high-sensitivity modified Glasgow prognostic score

INTERVENTIONS:
Other: Measurement of body composition with computed tomography (CT) — The cross section of the third lumbar vertebrae in the CT scan images of the patients will be analyzed for assessment of body composition parameters including skeletal muscle area (SMA), muscle radiation attenuation (MRA), visceral adipose tissue (VAT), subcutaneous adipose tissue (SAT)
  Groups: Subgroup of patients with available preoperative CT/MRI scans
Diagnostic Test: GLIM malnutrition criteria — GLIM criteria (Global Leadership Initiative on Malnutrition) will be applied to assess malnutrition
Diagnostic Test: EWGSOP2 sarcopenia criteria — EWGSOP2 criteria (Writing Group for the European Working Group on Sarcopenia in Older People 2) will be followed to determine the diagnosis of sarcopenia
  Groups: Subgroup of patients with available preoperative CT/MRI scans
Diagnostic Test: ESPEN-EASO criteria for sarcopenic obesity — The European Society for Clinical Nutrition and Metabolism (ESPEN) and the European Association for the Study of Obesity (EASO) consensus criteria from 2018 will be applied to assess sarcopenic obesity
  Groups: Subgroup of patients with available preoperative CT/MRI scans
Diagnostic Test: Prognostic Nutritional Index (PNI) — Prognostic Nutritional Index is diagnostic test based on serum albumin level and total lymphocyte count
Diagnostic Test: The high-sensitivity modified Glasgow prognostic score — The high-sensitivity modified Glasgow prognostic score (Hs-mGPS) is an inflammation-based score consisted of C-reactive protein level and serum albumin

SUMMARY:
This is a retrospective, observational study in consecutive patients operated on for primary RPS in the Institute of Oncology Ljubljana (Slovenia) between September 1999 and June 2020. This study aims to investigate the impact of preoperatively assessed body composition parameters on the perioperative outcomes of patients operated on for primary RPS. The impact of preoperative malnutrition, sarcopenia, sarcopenic obesity and myosteatosis to the oncologic and postoperative outcome in patients operated on for primary RPS will be examined. Additionally, the aim is to evaluate the prognostic role of preoperative immune and inflammatory markers (serum albumin level, C-reactive protein, neutrophil to lymphocyte ratio, platelet to lymphocyte ratio, high-sensitivity modified Glasgow prognostic score) and prognostic nutritional index in primary RPS patients undergoing surgery. Patient outcome will be evaluated in terms of overall survival (OS), local-recurrence free survival (LRFS), postoperative intrahospital length of stay, overall and major postoperative morbidity.

DETAILED DESCRIPTION:
Retroperitoneal sarcomas (RPS) are rare neoplasms of mesenchymal origin with estimated crude incidence of 0.3 cases per 100000 inhabitants per year. The most common histologic subtypes are well-differentiated and dedifferentiated liposarcoma and leiomyosarcoma, accounting for 42% and 26% of cases, respectively. RPS are optimally managed in multidisciplinary settings in specialized sarcoma centers. Surgical resection with an adequate margin of normal tissue is the cornerstone of curative therapy and en bloc surgical resection of localized tumors is the recommended surgical approach. This "extended" surgical approach (including resection of adjacent organs), is optimal for reducing local recurrence and improving overall survival.

Cancer patients undergoing surgical treatment face number of challenges which negatively impact their nutritional status. Patients are usually in catabolic state, which together with ongoing proteolysis and lipolysis as well as decreased protein synthesis contribute to development of cancer - associated cachexia. Most important nutritional disorders in these patients are malnutrition, sarcopenia, cancer cachexia. On the other side, often under-recognized, sarcopenic obesity is gaining attention in clinical and research settings.

The association of malnutrition and poor postoperative outcome has been demonstrated in patients with various cancer locations. Malnourished patients reportedly have longer length of postoperative stay (LOS), higher rates of 30-day mortality, infection rate, sepsis, reoperation, increased number of cardiopulmonary complications. Diagnostic process of malnutrition has been a topic of debate considering inconsistency in diagnostic methodology and criteria. Global Leadership Initiative on Malnutrition (GLIM) addressed this problem and recommended a new diagnostic scheme for malnutrition, in form of consensus report incorporating previous finding and recommendations from world leading clinical nutrition societies. To our knowledge, no study validated GLIM criteria in patients with primary RPS.

Sarcopenia is clinical syndrome characterized by generalized skeletal muscle mass loss, loss of strength and function (performance). Sarcopenia has been associated with lower survival rate and proved to be an independent predictor of survival in patients with breast cancer, pancreatic adenocarcinoma, hepatocellular carcinoma, and melanoma. There is a lack of studies investigating the impact of sarcopenia on survival and postoperative outcome in patients with soft-tissue sarcoma (STS), including retroperitoneal sarcoma. Similarly to malnutrition diagnosis, there is an evident inconsistency and confusion in diagnostic criteria and tools used to define and characterize sarcopenia in clinical practice and research. However, recently the European Working Group on Sarcopenia in Older People (EWGSOP2) published updated findings in form of Revised European Consensus. The Working Group proposed new recommendation, among which are those related to establishing specific cut-off points for body composition (primarily skeletal muscle quantity and quality) measures that identify and characterize sarcopenia.

Sarcopenic obesity (SO) is co-existence of sarcopenia and excess adiposity. Recent expert consensus of The European Society for Clinical Nutrition and Metabolism (ESPEN) and the European Association for the Study of Obesity (EASO) will be followed for definition and diagnostic criteria for SO.

Myosteatosis is ectopic adipose tissue infiltration in skeletal muscle. Intermuscular adipose tissue can be quantified using CT scans by low muscle radiodensity. CT-derived myosteatosis contributes to impaired glucose metabolism, including insulin resistance, type 2 diabetes mellitus, and inflammation. Additionally, it may increase the risk for dyslipidemia. Myosteatosis may predict oncologic and postoperative outcome in primary RPS patients.

Patients with primary RPS are in a great risk for malnutrition, sarcopenia and cachexia for the number of reasons: requirement for demanding abdominal surgery in their management, catabolic tumor effects, long period before diagnosis of RPS and tumor size (approximately 15 cm). Due to their rarity, it is still unclear how preoperative nutritional status and body composition impact outcome of patients with primary RPS.

STUDY DESIGN DATA COLLECTION Patient's histories including the anaesthetician's preoperative reports, surgeon's operative reports, hospital records, and follow-up data will be collected. Paper and electronic data archive of Institute of Oncology Ljubljana Patient Data Information System will be used.

The following preoperative clinical data will be acquired: age, sex, preoperative weight, height, significant weight loss, appetite loss and weakness. CT reports will be also acquired for analysis as well as histopathological diagnosis (subtype), stage, grade and tumor size.

The preoperative laboratory data, including absolute counts of leukocytes, neutrophils, lymphocytes, monocytes and platelets, CRP, and albumin levels will be assessed. Data will be deidentified and whenever possible all measures to conceal patient identifiers and maintain patient confidentiality will be taken.

STATISTICAL CONSIDERATIONS The data will be presented using appropriate summary statistics: mean, median, standard deviation for continuous variables and percentages and frequencies for categorical variables. Kaplan-Meier method will be used for survival curves analysis and differences between survival rates compared using the log-rank test. The independent prognostic variables for survival (OS and LRFS) will be identified using Cox proportional hazard model (hazard ratio, 95% confidence interval, p value).

ETHICS The study was approved by Slovenian National Medical Ethics Committee, Institute of Oncology Ljubljana Review Board and Institute of Oncology Ljubljana Ethical Committee. The need to obtain informed consent from participants was waived.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged above 18 years old
* Patients with primary localized RPS or pelvic sarcoma operated at Surgical Department of Institute of Oncology in Ljubljana

Exclusion Criteria:

* Patients with Gastrointestinal Stromal Tumors (GISTs) and Retroperitoneal desmoid-type fibromatosis (DF)
* Patients with visceral sarcomas (arising from visceral organ i.e., gastrointestinal, and genitourinary tracts sarcoma)
* Patients with benign retroperitoneal / pelvic tumors
* Patients with residual RPS operated at another hospital
* Patients with present recurrent, secondary, and metastatic RPS
* Unable to access patients' data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients operated on for primary RPS in the Institute of Oncology Ljubljana (Slovenia) between September 1999 and June 2020
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | within 30 days after surgery
  Complications graded by Clavien-Dindo Complication Classification System
Local recurrence rate | From date of surgery until the date of first documented local progression assessed until June 2020
  A postoperative local recurrence will be defined by biopsy-proven or radiographic evidence of local recurrent disease
Mortality | Length of survival after surgery until June 2020 (up to 130 months)
  Overall survival (OS) will be defined as the time between the date of the operation to the date of death from any cause or last follow-up (according to medical records and using telephone contacts)

SECONDARY OUTCOMES:
Length of hospital stay | up to 90 days after surgery
  Time interval from the date of operation to the date of discharge. Body composition parameters may predict the length of hospital stay
Major postoperative morbidity | within 90 days after surgery
  Complication grade 3 or higher according to Clavien-Dindo Complication Classification System
Prevalence of preoperative malnutrition in primary RPS patients | within 30 days before surgery
  A prevalent case of malnutrition will be considered if a patient fulfills the Global Leadership Initiative on Malnutrition (GLIM) criteria. GLIM proposed 5 diagnostic criteria to assess malnutrition and includes 3 phenotypic (weight loss, low body mass index and reduced muscle mass) and 2 etiologic (reduced food intake/assimilation, and inflammation/disease burden) criteria. To diagnose malnutrition at least 1 phenotypic criterion and 1 etiologic criterion should be present
Prevalence of preoperative sarcopenia in primary RPS patients | within 30 days before surgery
  A prevalent case of sarcopenia will be considered if a patient fulfills the diagnostic criteria defined by European Working Group on Sarcopenia in Older People (EWGSOP2)
To evaluate the impact of skeletal muscle area (SMA) on the prognosis of patients with primary RPS | through study completion, an average of 6 months
  Skeletal muscle area (SMA) area will be measured by using preoperative computed tomography (CT) scans at lumbar (L3) vertebral level and recorded as cm^2 using standard Hounsfield Unit thresholds of - 29 to + 150. SMA at the third lumbar spine level has been established as a good indicator of whole-body muscle mass.
To evaluate the impact of the muscle radiation attenuation (MRA) on the prognosis of patients with primary RPS | through study completion, an average of 6 months
  Muscle radiation attenuation (MRA) will be assessed using CT scans at lumbar (L3) vertebral level and recorded as mean Hounsfield unit (HU) of each pixel within a region of interest. MRA reflects muscle composition, including the degree of intramuscular fat accumulation, important to define the presence of myosteatosis
To evaluate the impact of visceral adipose tissue (VAT) on the prognosis of patients with primary RPS | through study completion, an average of 6 months
  Visceral adipose tissue (VAT) area will be measured by using preoperative computed tomography (CT) scans at lumbar (L3) vertebral level and recorded as cm^2 using standard Hounsfield Unit thresholds of -150 to -50
To evaluate the impact of subcutaneous adipose tissue (SAT) on the prognosis of patients with primary RPS | through study completion, an average of 6 months
  Subcutaneous adipose tissue (SAT) area will be measured by using preoperative computed tomography (CT) scans at lumbar (L3) vertebral level and recorded as cm^2 using standard Hounsfield Unit thresholds of -190 to -30.
To evaluate the impact of visceral-to-subcutaneous adipose tissue area ratio (VSR) on the prognosis of patients with primary RPS | through study completion, an average of 6 months
  Visceral-to-subcutaneous adipose tissue ratio will be calculated by dividing the visceral adipose tissue area by the subcutaneous adipose tissue area.
To assess the impact of complete blood count based systemic inflammatory markers: NLR, PLR and SII on the prognosis of patients with primary RPS | within 30 days before surgery
  Neutrophil to lymphocyte ratio (NLR): calculated as the absolute neutrophil count divided by the absolute lymphocyte count.
  Platelet to Lymphocyte Ratio (PLR): calculated as the absolute platelet count divided by the absolute lymphocyte count.
  Systemic immune inflammation index (SII): based on absolute platelet, neutrophil and lymphocyte count and calculated according to following formula:
  SII =(platelet count×neutrophil count)/(lymphocyte count)
To assess the preoperative high-sensitivity modified Glasgow prognostic score (Hs-mGPS) and prognostic nutrition index (PNI) as prognostic tools in primary RPS patients | within 30 days before surgery
  The high-sensitivity modified Glasgow prognostic score (Hs-mGPS) will be defined as numeric value 0 - 2 according to following criteria based on C-reactive protein (CRP) and serum albumin levels:
  Score 0: CRP level ≤ 0.3 mg/dl and albumin ≥ 3.5 g/dl, Score 1: CRP level > 0.3 mg/dl and albumin ≥ 3.5 g/dl, Score 3: CRP level > 0.3 mg/ dl and albumin < 3.5 g/dl.
  The prognostic nutrition index (PNI) will be calculated based on previously published and validated formula:
  PNI =10× serum albumin (g/dl)+0.005× lymphocyte count (per mm^3)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Ramanović, M.D., Principal Investigator — Institute of Oncology Ljubljana, Ljubljana
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided
Not decided

REFERENCES:
- [Background] Previtali P, Fiore M, Colombo J, Arendar I, Fumagalli L, Pizzocri M, Colombo C, Rampello NN, Mariani L, Gronchi A, Codazzi D. Malnutrition and Perioperative Nutritional Support in Retroperitoneal Sarcoma Patients: Results from a Prospective Study. Ann Surg Oncol. 2020 Jun;27(6):2025-2032. doi: 10.1245/s10434-019-08121-0. Epub 2019 Dec 17. PMID 31848820
- [Background] Stiller CA, Trama A, Serraino D, Rossi S, Navarro C, Chirlaque MD, Casali PG; RARECARE Working Group. Descriptive epidemiology of sarcomas in Europe: report from the RARECARE project. Eur J Cancer. 2013 Feb;49(3):684-95. doi: 10.1016/j.ejca.2012.09.011. Epub 2012 Oct 15. PMID 23079473
- [Background] Arends J, Baracos V, Bertz H, Bozzetti F, Calder PC, Deutz NEP, Erickson N, Laviano A, Lisanti MP, Lobo DN, McMillan DC, Muscaritoli M, Ockenga J, Pirlich M, Strasser F, de van der Schueren M, Van Gossum A, Vaupel P, Weimann A. ESPEN expert group recommendations for action against cancer-related malnutrition. Clin Nutr. 2017 Oct;36(5):1187-1196. doi: 10.1016/j.clnu.2017.06.017. Epub 2017 Jun 23. PMID 28689670
- [Background] Cederholm T, Jensen GL, Correia MITD, Gonzalez MC, Fukushima R, Higashiguchi T, Baptista G, Barazzoni R, Blaauw R, Coats A, Crivelli A, Evans DC, Gramlich L, Fuchs-Tarlovsky V, Keller H, Llido L, Malone A, Mogensen KM, Morley JE, Muscaritoli M, Nyulasi I, Pirlich M, Pisprasert V, de van der Schueren MAE, Siltharm S, Singer P, Tappenden K, Velasco N, Waitzberg D, Yamwong P, Yu J, Van Gossum A, Compher C; GLIM Core Leadership Committee; GLIM Working Group. GLIM criteria for the diagnosis of malnutrition - A consensus report from the global clinical nutrition community. Clin Nutr. 2019 Feb;38(1):1-9. doi: 10.1016/j.clnu.2018.08.002. Epub 2018 Sep 3. PMID 30181091
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Donini LM, Busetto L, Bischoff SC, Cederholm T, Ballesteros-Pomar MD, Batsis JA, Bauer JM, Boirie Y, Cruz-Jentoft AJ, Dicker D, Frara S, Fruhbeck G, Genton L, Gepner Y, Giustina A, Gonzalez MC, Han HS, Heymsfield SB, Higashiguchi T, Laviano A, Lenzi A, Nyulasi I, Parrinello E, Poggiogalle E, Prado CM, Salvador J, Rolland Y, Santini F, Serlie MJ, Shi H, Sieber CC, Siervo M, Vettor R, Villareal DT, Volkert D, Yu J, Zamboni M, Barazzoni R. Definition and Diagnostic Criteria for Sarcopenic Obesity: ESPEN and EASO Consensus Statement. Obes Facts. 2022;15(3):321-335. doi: 10.1159/000521241. Epub 2022 Feb 23. PMID 35196654
- [Background] Hou T, Guo T, Nie R, Hong D, Zhou Z, Zhang X, Liang Y. The prognostic role of the preoperative systemic immune-inflammation index and high-sensitivity modified Glasgow prognostic score in patients after radical operation for soft tissue sarcoma. Eur J Surg Oncol. 2020 Aug;46(8):1496-1502. doi: 10.1016/j.ejso.2020.05.026. Epub 2020 Jun 11. PMID 32576479
- [Background] Yang Z, Zhang B, Hou L, Xie Y, Cao X. Pre-operative prognostic nutritional index predicts the outcomes for triple-negative breast cancer. Tumour Biol. 2014 Dec;35(12):12165-71. doi: 10.1007/s13277-014-2524-6. Epub 2014 Aug 30. PMID 25172099